CLINICAL TRIAL: NCT06500013
Title: Intervention With WhatsApp Messaging to Assess the Effect of Self-designed Messages and Standardized Messages in Adherence to Antiretroviral Treatment in Young People Living With HIV in a Hospital in Lima, Peru: Randomized Control Trial
Brief Title: WhatsApp Intervention to Assess the Effect of Messages in Adherence to Antiretrovirals in Young People With HIV in Peru
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Principal Investigator, Jeffrey Freidenson, Principal Investigator, Universidad Peruana Cayetano Heredia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 104475
Record Dates: First submitted 2024-06-29; First posted 2024-07-15 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: HIV
Keywords: HIV; mHealth; messages; adherence; ART; antiretroviral therapy

STUDY DESIGN:
Intervention Model Description: Parallel model with 1:1 assignment to one of two study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-designed messages (Experimental): This group of participants will design their own messages, and receive them via mobile messaging up to 3 times a week in the day and time of their choosing, for 16 weeks.
  Interventions: Behavioral: Self-designed messages
- Standardized messages (Active Comparator): This group of participants will receive messages designed by researchers based on behavioral change theories, up to 3 times a week in the day and time of their choosing, for 16 weeks.
  Interventions: Behavioral: Standardized messages

INTERVENTIONS:
Behavioral: Self-designed messages — Messages designed by participants
  Arms: Self-designed messages
Behavioral: Standardized messages — Messages designed by researchers based on behavioral change theories
  Arms: Standardized messages

SUMMARY:
The goal of this clinical trial is to learn which type of messages is more efficacious to improve adherence to medication in young people living with HIV. The main question is aims to answer is:

-Are messages designed by participants (self-designed) more efficacious than messages designed by health providers to improve adherence to antiretroviral treatment (HIV medications)?

Researchers will compare both types of messages to see if one is better than the other in helping participants take their medications.

Participants will:

* Receive either messages designed by themselves or by health providers for 4 months.
* Be able to chat with health providers at any time, with special focus regarding questions about their condition, medications and health services.
* Complete questionnaires via WhatsApp describing how they are taking their medications, and how often they forget to take them.
* Complete questionnaires via WhatsApp describing their opinion about receiving the messages and being able to chat with health providers.

ELIGIBILITY:
Inclusion Criteria:

* People living with HIV of age 18-29 at the moment of signing informed consent.
* Being a patient of the study center's Infectious Diseases clinic or National HIV Program, between March 2024 and July 2024.
* Ownership of a mobile phone that supports WhatsApp.

Exclusion Criteria:

* Being pregnant at the moment of signing informed consent.
* Being illiterate at the moment of signing informed consent.
* Being blind at the moment of signing informed consent

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — * Male
  * Female
  * Transgender
  * Other
Enrollment: 131 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Result of SMAQ Questionnaire Adjusted for the Effect of Covariables | Baseline, 16 weeks.
  The SMAQ questionnaire evaluates medication adherence. It provides a dichotomic result of adherence (yes/no), and a semiquantitative estimate of adherence. Greater than 95% adherence is considered as adherent, and less than 95% as non-adherent.

SECONDARY OUTCOMES:
ART adherence measured by SMAQ Questionnaire at 4, 8 and 12 weeks of intervention | 4, 8 and 12 weeks of intervention
  SMAQ provides a dichotomic result of adherence (yes/no): we will report percentage of participants adherent to ART per study group during the intervention.
Loss to follow-up | From the start of delivery intervention until study completion
  Loss to follow-up is defined as either (i) participants not responding to messages for ≥ 30 continuous days since receiving the intervention and not responding to messages or questionnaires at the end of their intervention period (t=16), or (ii) particip
Time of permanence in the study | Baseline until study completion (16 weeks).
  Time of permanence in the study, indicated from the first date of intervention delivery until loss to-follow up or study completion. We will describe the median and interquartile range of this result in both study arms.
Metrics on the use of a bidirectional platform for intervention delivery | End of the intervention at 16 weeks.
  Frequencies, percentages, and means with a standard deviation of messages and questionnaires programmed for sending, sent, received, read, and answered by participants. Frequencies and percentages of different process indicators self-reported by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Freidenson, M.D, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (1):
- Hospital Cayetano Heredia, Lima, Lima Province, Peru

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data collected during the trial will be made available 6 months after study completion. Access will be provided after a formal request has been reviewed and approved by the Institutional Review Boards of the study sponsor and study center, and with a signed data sharing agreement. The study protocol, informed consent, and statistical analysis plan will be published in a peer-reviewed journal. Requested data and clinical study reports will be provided through a secure data-sharing platform.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 6 months after the trial ends, until 5 years after the trial end date.
Access Criteria: IPD may be shared to qualified researchers for scientific purposes. This will require the review and approval of a formal petition including the research proposal and statistical analysis plan, and a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Freidenson-Bejar J, Espinoza D, Calderon-Flores R, Mejia F, Gonzalez-Lagos E. Intervention With WhatsApp Messaging to Compare the Effect of Self-Designed Messages and Standardized Messages in Adherence to Antiretroviral Treatment in Young People Living With HIV in a Hospital in Lima, Peru: Protocol for a Nonblinded Randomized Controlled Trial. JMIR Res Protoc. 2025 May 22;14:e66941. doi: 10.2196/66941. PMID 40403302